CLINICAL TRIAL: NCT01015014
Title: First-in-human, Two-stage, Randomized, Placebo-controlled, Double-blind, Dose Escalation Study To Determine The Safety, Tolerability, And Pharmacokinetic Profile Of An3365 In Single And Multiple Doses In Young Healthy Subjects
Brief Title: Safety, Pharmacokinetics (PK) and Tolerability Study of a Novel Drug for Treatment of Bacterial Infections
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AN3365-PK-101; C3501001 (Other: Alias Study Number)
Record Dates: First submitted 2009-10-20; First posted 2009-11-17 (Estimated); Last update posted 2019-03-05 (Actual); Status verified 2019-03

CONDITIONS: Gram-negative Bacterial Infection
Keywords: Gram negative; bacteria; infection
MeSH Terms: conditions — Gram-Negative Bacterial Infections; Infections

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- AN3365 (Active Comparator)
  Interventions: Drug: AN3365
- Saline (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AN3365 — LP, 600 mg vial; reconstituted in Normal Saline
  Arms: AN3365
Drug: Placebo — 0.9% sodium chloride for injection
  Arms: Saline

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability and pharmacokinetic profile of an antibacterial compound for treatment of hospital acquired Gram negative infection.

DETAILED DESCRIPTION:
Single-center, randomized, placebo-controlled, double-blind study to determine the safety, tolerability and pharmacokinetic profile of compound in single and multiple doses in young healthy males.

ELIGIBILITY:
Inclusion Criteria:

* Young healthy males, 18-45 years (inclusive) of age
* Healthy as judged by a responsible physician with no clinically significant abnormality
* Surgically sterile OR agrees to abstain from sexual intercourse with a female partner OR agrees to use a condom and spermicide during sexual intercourse with a female partner who uses another form of contraception
* Body weight above 50 kg (Body Mass Index between 19 and 30 kg/m2)
* Non-smokers
* Willing and able to comply with study instructions and commit to all follow-up visits
* Ability to understand, agree to and sign the study Informed Consent Form (ICF)

Exclusion Criteria:

* History of serious adverse reactions or hypersensitivity to any drug; or who have a known allergy to any of the test product(s) or any components in the test product(s); or history of hypersensitivity or allergic reactions to any of the study preparations as described in the Investigator's Brochure
* Any clinically significant central nervous system, cardiac, pulmonary, metabolic, renal, hepatic or gastrointestinal conditions
* Abnormal physical findings of clinical significance at the screening examination or baseline
* History of orthostatic hypotension
* Clinically significant abnormal laboratory values
* Presence or history of allergies requiring acute or chronic treatment
* 12 lead ECG abnormalities
* Major surgical interventions within 6 months of the study
* Has a positive pre-study Hepatitis B surface antigen; positive hepatitis C (HCV) antibody or detectable HCV ribonucleic acid (RNA); or positive HIV antibody result
* Use of prescription or non-prescription drugs
* Has a history of regular alcohol consumption
* Loss of 500 mL blood or more during the 3 month period before the study
* People that follow vegetarian or vegan diet
* Symptoms of a significant somatic or mental illness in the four week period preceding drug administration
* History of drug abuse or dependence within 12 months of the study
* The subject has a positive pre-study alcohol or urine drug screen
* Concurrent participation in another drug or device research study or within 60 days of post participation in another drug or device study
* Considered by the Investigator to be unsuitable candidate for this study

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 64 (Actual)
Dates: Start 2009-11-05 (Actual); Primary Completion 2010-05-13 (Actual); Study Completion 2010-05-13 (Actual)

PRIMARY OUTCOMES:
Clinical safety data from 12-lead ECG, clinical laboratory tests, urinalysis, injection site tolerability, spontaneous/elicited adverse event reporting, and vital signs (blood pressure, heart rate, respiratory rate) | Multiple time points up to 14 days

SECONDARY OUTCOMES:
Assessment of pharmacokinetic parameters to achieve appropriate exposure and estimate the dose proportionality | Multiple time points up to 14 days

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- CMAX, Adelaide, Australia